CLINICAL TRIAL: NCT01441193
Title: A Phase I, Open Label, Safety and Immunogenicity Vaccine Trial Based on the Association of Recombinant HIV-1 Biologically Active Tat and V2-deleted Env Proteins in HIV Uninfected Healthy Adult Volunteers.
Brief Title: A Phase I Safety and Immunogenicity Preventive Vaccine Trial Based on the HIV-1 Tat and V2-deleted Env Proteins (ISS P-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollments were suspended due to delta-V2 Env unavailability, following the EMA/CHMP/BWP/534898/2008 guideline, not allowing the use of a retest date
Sponsor: Barbara Ensoli, MD (Other)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ISS P-002
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infection
Keywords: HIV; preventive vaccine; Tat; Env
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HIV-1 Tat/delta-V2 Env combined vaccine (Experimental): Tat 7.5 microg and delta-V2 Env 100 microg associated proteins administered i.d. (priming) at week 0, 4 and 8 or i.m. (boosting) at weeks 24 and 36
  Interventions: Biological: HIV-1 Tat/delta-V2 Env combined vaccine
- HIV-1 delta-V2 Env vaccine (Active Comparator): delta-V2 Env 100 microg administered i.d. (priming) at week 0, 4 and 8 or i.m. (boosting) at week 24 and 36
  Interventions: Biological: HIV-1 delta-V2 Env vaccine
- HIV-1 Tat vaccine 7.5 microg (Active Comparator): Tat 7.5 microg administered i.d. (priming) at week 0, 4 and 8 or i.m. (boosting) at week 24 and 36
  Interventions: Biological: HIV-1 Tat vaccine 7.5 microg
- HIV-1 Tat vaccine 30 microg (Active Comparator): Tat 30 microg administered i.d. at week 0, 4 and 8
  Interventions: Biological: HIV-1 Tat vaccine 30 microg

INTERVENTIONS:
Biological: HIV-1 Tat/delta-V2 Env combined vaccine
  Arms: HIV-1 Tat/delta-V2 Env combined vaccine
Biological: HIV-1 delta-V2 Env vaccine
  Arms: HIV-1 delta-V2 Env vaccine
Biological: HIV-1 Tat vaccine 7.5 microg
  Arms: HIV-1 Tat vaccine 7.5 microg
Biological: HIV-1 Tat vaccine 30 microg
  Arms: HIV-1 Tat vaccine 30 microg

SUMMARY:
This Phase I study was directed at evaluating the safety profile and the immunogenicity of the vaccination with recombinant HIV-1 Tat and V2-deleted Env (delta-V2 Env) proteins administered in association in healthy, immunologically competent adults, compared to delta-V2 Env or Tat alone.

DETAILED DESCRIPTION:
Since the inexorable spreading of HIV pandemic is unabated, the urgency of designing an effective, safe, inexpensive and easily administrable vaccine to protect people from HIV and/or AIDS is an absolute priority. Considering the array of functions sequentially exerted by the regulatory and the structural gene products in supporting the setting of a primary HIV infection, it is expected that vaccines combining early and late viral products (combined vaccines) should be superior to the single antigens approaches since they target multiple viral proteins which are necessary at different key steps of the virus life cycle, including cell-to-cell virus transmission and systemic virus propagation. A combined vaccine strategy based on the early regulatory protein Tat in association with the late structural protein Env modified to increase its immunogenicity (delta-V2Env) has been evaluated in pre-clinical studies in both small animals and monkeys. The results of these studies indicated that the combination of Tat with delta-V2Env is superior in inducing specific immune responses against both Tat and delta-V2Env antigens and in protecting or containing virus replication more efficiently than vaccination with the single antigens alone, confirming that these proteins represent optimal co-antigens for a combined vaccine strategy.

This study was a multicentric, open label, randomized phase I trial, directed to qualify the safety and the immunogenicity of the vaccine based on the association of HIV-1 biologically active Tat and oligomeric ΔV2 Env proteins in healthy, immunologically competent adult volunteers, compared to the single compounds. Tat and delta-V2 Env proteins either in association or as single compounds were administered by a prime-boost regimen, consisting of 3 intradermal priming doses followed by 2 intramuscular boosting injections. Of note, phase I trials have already been successfully conducted with the 2 single components, at the doses proposed in this trial, in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years;
2. Negative blood pregnancy test for women of childbearing potential at screening evaluation (a urine dipstick test will be repeated just before each vaccination), and use of an acceptable mean of contraception by both men and women, since one month prior to immunization (only for women) and until at least 6 months after the last immunization;
3. Blood pressure, heart rate and ECG within normal ranges or with mild alterations acknowledged as non clinically significant by the site clinician;
4. Haematological and biochemical parameters within the clinical site normal ranges or with mild alterations acknowledged by the site clinician as non clinically significant;
5. Normal urine dipstick with esterase and nitrite;
6. Normal thyroid function;
7. Negative for HIV infection and for anti-Tat antibodies;
8. Good physical and mental health status;
9. Availability for the planned study duration;
10. Signed informed consent.

Exclusion Criteria:

1. Concomitant neoplastic diseases;
2. History of malignant neoplastic diseases;
3. History of encephalopathy, neuropathy or unstable CNS pathology, immunodeficiency, autoimmune disease, angina or cardiac arrhythmias, or any other clinically significant medical problems;
4. History of anaphylaxis or serious adverse reactions to vaccines as well as serum IgE levels exceeding 1,000 U.I./mL;
5. History of serious allergic reaction to any substance, requiring hospitalization or emergency medical care;
6. Chest radiography showing evidence of active or acute cardiac or pulmonary disease;
7. Any unstable cardiovascular disease;
8. Active syphilis by TPHA and RPR tests [NOTE: If the serology is documented to be a false positive or due to an adequately treated infection, the volunteer is eligible];
9. Active tuberculosis by cutaneous TB diagnostic test [NOTE: Volunteers with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring specific therapy are eligible];
10. Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol. Persons with psychotic disorders, major affective disorders or suicidal ideation are specifically excluded;
11. Current use of psychotropic drugs;
12. Drug and/or alcohol abuse;
13. Current or prior therapy with immunomodulators or immunosuppressive drugs and anticoagulant drugs within 30 days prior to study medication administration;
14. Live attenuated vaccines within 60 days prior to study entry [NOTE: Medically indicated sub-unit or killed vaccines (e.g, influenza, pneumococcal, hepatitis A and B) are not exclusionary, but should be given at least 4 weeks away from anti-HIV immunizations];
15. Use of investigational agents within 90 days prior to study entry;
16. Participation in another experimental protocol within 6 months prior to pre-study screening;
17. Prior receipt of HIV vaccine in a previous HIV vaccine trial;
18. Receipt of blood products or immunoglobulin in the past 6 months;
19. Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity | up to week 68
  To qualify the vaccine candidate as safe and immunogenic by evaluating the number of local and systemic adverse events, including any significant change in hematological/biochemical/coagulation laboratory parameters, and the frequency of anti-Tat and anti-delta-V2 Env humoral and cellular immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, Study Director — Istituto Superiore di Sanità
Locations (3):
- Italy (3):
  - Policlinico di Modena, Divisione di Malattie Infettive, Modena
  - Azienda Ospedaliera San Gerardo, Divisione di Malattie Infettive, Monza
  - IFO - S. Gallicano, Dermatologia Infettiva, Rome

REFERENCES:
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Caputo A, Gavioli R, Bellino S, Longo O, Tripiciano A, Francavilla V, Sgadari C, Paniccia G, Titti F, Cafaro A, Ferrantelli F, Monini P, Ensoli F, Ensoli B. HIV-1 Tat-based vaccines: an overview and perspectives in the field of HIV/AIDS vaccine development. Int Rev Immunol. 2009;28(5):285-334. doi: 10.1080/08830180903013026. PMID 19811313
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Barnett SW, Srivastava IK, Ulmer JB, Donnelly JJ, Rappuoli R. Development of V2-deleted trimeric envelope vaccine candidates from human immunodeficiency virus type 1 (HIV-1) subtypes B and C. Microbes Infect. 2005 Nov;7(14):1386-91. doi: 10.1016/j.micinf.2005.07.018. Epub 2005 Sep 20. PMID 16275150
- [Background] Ensoli B, Cafaro A, Caputo A, Fiorelli V, Ensoli F, Gavioli R, Ferrantelli F, Cara A, Titti F, Magnani M. Vaccines based on the native HIV Tat protein and on the combination of Tat and the structural HIV protein variant DeltaV2 Env. Microbes Infect. 2005 Nov;7(14):1392-9. doi: 10.1016/j.micinf.2005.07.016. Epub 2005 Sep 15. PMID 16243561
- [Background] Caputo A, Brocca-Cofano E, Castaldello A, Voltan R, Gavioli R, Srivastava IK, Barnett SW, Cafaro A, Ensoli B. Characterization of immune responses elicited in mice by intranasal co-immunization with HIV-1 Tat, gp140 DeltaV2Env and/or SIV Gag proteins and the nontoxicogenic heat-labile Escherichia coli enterotoxin. Vaccine. 2008 Feb 26;26(9):1214-27. doi: 10.1016/j.vaccine.2007.12.030. Epub 2008 Jan 15. PMID 18243435
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- See also: Click here for a description of the efforts by the Italian National AIDS Center at the Italian National Institute of Health to develop preventive and therapeutic HIV vaccines based on the HIV-1 Tat protein — http://www.hiv1tat-vaccines.info